CLINICAL TRIAL: NCT03822585
Title: Detection of β-thalassemia Carriers Among Close Relatives of β-thalassemia Children Attending Assiut University Children Hospital
Brief Title: Detection Of β-thalassemia Carriers In Assiut
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Mohammed Radi Abdelhakeem, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Thalassemia Carriers
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Beta-Thalassemia
Keywords: HbA2, HPLC
MeSH Terms: conditions — beta-Thalassemia | interventions — Blood Cell Count

STUDY DESIGN:
Intervention Model Description: Close Relatives Of β-Thalassemia Will Do Laboratory Tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Close Relatives Of β-thalassemia (Other): Laboratory diagnostic tests as (CBC, Iron Study, Serum Ferritin, HPLC, Genetic study) will be done to Brothers, Sisters & Cousins of β-thalassemia Children With Microcytic Hypochromic Anemia Attending Assiut University Child Hospital
  Interventions: Diagnostic Test: CBC, Iron Study, Serum Ferrittin, HPLC,Genitic Study

INTERVENTIONS:
Diagnostic Test: CBC, Iron Study, Serum Ferrittin, HPLC,Genitic Study — high performance liquid chromatography (HPLC) has become the preferred technique, as it can detect most of the clinically significant variants. polymerase chain reaction (PCR)-based procedures detect Commonly occurring mutations of the HBB gene .
  If targeted mutation analysis fails to detect the mutation, scanning or sequence analysis can be used. Sensitivity of both mutation scanning and sequence analysis is 99%.

SUMMARY:
Thalassemia is different in kids with microcytic hypochromic anemia than general population because there is a confusion between symptoms of thalassemia and iron deficiency anemia in kids and both of them differ in management and prognosis. otherwise the most commonest causes of microcytic hypochromic anemia in kids are iron deficiency anemia and thalassemia and both of them are more common in kids than in general population.

Thalassemia is different in Egypt than anywhere in the world because there is no accurate estimation of incidence and prevalence of such dangerous disease in Egypt inspite of many cases attending thalassemia center (hundreds) and this disease is autosomal recessive and its incidence can be minimized by detection of carrier cases by gene study hopping that to be done as a routine premarital investigation.

DETAILED DESCRIPTION:
The term "thalassemia" is derived from the Greek words "Thalassa"(sea) and "Haema" (blood) and refers to disorder associated with defective synthesis of α or β-globin subunits of haemoglobin HbA

There are two main types of thalassemia:

α-thalassemia is one of the most common hemoglobin genetic abnormalities and is caused by the reduced or absent production of the alpha globin chains. Alpha-thalassemia is prevalent in tropical and subtropical world regions where malaria was and still is epidemic, but as a consequence of the recent massive population migrations, alpha-thalassemia has become a relatively common clinical problem in North America, North Europe, and Australia

β-thalassemia syndromes are a group of hereditary blood disorders characterized by reduced or absent beta globin chain synthesis, resulting in reduced Hb in red blood cells (RBC), decreased RBC production and anemia. Most thalassemias are inherited as recessive traits. The phenotypes of homozygous or genetic heterozygous compound β-thalassemias include thalassemia major and thalassemia intermedia. Individuals with thalassemia major usually come for medical attention within the first two years of life and require regular RBC transfusions to survive. Thalassemia intermedia include patients who present later and do not require regular transfusion. Except in the rare dominant forms, heterozygous β-thalassemia results in the clinically silent carrier state. HbE/ β-thalassemia and HbC/ β-thalassemia exhibit a great range in terms of diversity of phenotypes and spectrum of severity. People who are carriers of the disease received variant genes from one parent and normal gene from the other parent

Thalassemia is widespread throughout ,they are more prevalent in people living in South-East Asia, South Asia, Middle East, and Mediterranean regions

Thalassemia is the most common form of inherited anemia worldwide. The World Health Organization reports suggest that about 60,000 infants are born with a major thalassemia every year. Although individuals originating from the tropical belt are most at risk, it is a growing global health problem due to extensive population migrations

Population migration and intermarriage between different ethnic groups has introduced thalassemia in almost every country of the world

In Egypt, β -thalassemia is the most common type with a carrier rate varying from 5.3 to 9% and a gene frequency of 0.03. So, it was estimated that 1,000/1.5 million per year live births will suffer from thalassemia disease in Egypt (total live births 1,936,205 in 2006)

β Thalassemia creates a social and financial burden for the patients' family and the Egyptian government. The high frequency of beta-thalassemia carriers with increasing rate of newly born cases is a pressing reason for the importance to develop prevention program for beta-thalassemia in Egypt

The thalassaemia syndromes, particularly those requiring multiple blood transfusions, are a serious burden on health services and a problem which may be increasing on a global scale . Even milder syndromes, known as thalassaemia intermedia or non-transfusion dependent thalassaemia, require careful follow up since complications are expected over time in the natural course of the disease

The need for lifelong follow up and care and the occurrence of complications affecting major organs such as liver, heart and endocrine glands, creates the need for organised expert services and also the need for major resources in terms of essential drugs and donated blood for transfusions. In terms of clinical outcomes, The investigator expect that patients will survive with the best possible quality of life, if treated holistically in an expert centre

Detection of asymptomatic carriers by reliable laboratory methods is the cornerstone of prevention of this serious health problem. high performance liquid chromatography (HPLC) has become the preferred technique, as it can detect most of the clinically significant variants. The simplicity of the automated system with internal sample preparation, superior resolution, rapid assay time, and accurate quantification of hemoglobin fractions makes this an ideal methodology for the routine clinical laboratory

Commonly occurring mutations of the HBB gene are detected by a number of polymerase chain reaction (PCR)-based procedures. The most commonly used methods are reverse dot blot analysis or primer-specific amplification with a set of probes or primers complementary to the most common mutations in the population from which the affected individual originated

Other methods based on real-time PCR or microarray technology because of their reproducibility, rapidity, and easy handling are potentially suitable for the routine clinical laboratory

If targeted mutation analysis fails to detect the mutation, scanning or sequence analysis can be used. Sensitivity of both mutation scanning and sequence analysis is 99%. In the meantime, the presence of an extended deletion should be investigated by using multiplex ligation-dependent probe amplification (MPLA)

Screening for genetic diseases aims to reduce the burden of these disorders on individuals by identifying those at increased risk, thereby enabling individuals to receive information about personal health, future health and/or potential health of offspring

At risk individuals must be provided with information regarding the mode of inheritance, the genetic risk of having affected children and the natural history of the disease including the available treatment and therapies under investigation

Several countries have set up comprehensive national prevention programs, which include public awareness and education, carrier screening, and counseling, as well as information on prenatal diagnosis and preimplantation diagnosis. These countries are Italy, Greece, Cyprus, UK, France, Iran, Thailand, Australia, Singapore, Taiwan, Hong Kong, and Cuba

ELIGIBILITY:
Inclusion Criteria:

* Close Relatives Of B-Thalassemia Carriers With Microcytic Hypochromic Anemia

Exclusion Criteria:

* Normocytic Normochromic Anemia
* Iron Deficiency Anemia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
detection of thalassemia carriers in children with microcytic hypochromic anemia | 2 years
  accurate detection of prevalence rate of thalassemia carriers among relatives of β-thalassemia

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed HM Ghazally, PROF, Study Director — Assiut University Child Hospital

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will become available in January 2021 for unlimited years
Access Criteria: Through finding the research in the site of ClinicalTrials.gov
URL: http://shimaaradi2007@yahoo.com